CLINICAL TRIAL: NCT04207879
Title: Longitudinal Profiling of Gut Microbiome in Overweight or Obese Participants on a Modified Atkins Diet: a Prospective Cohort Study
Brief Title: Modified Atkins Diet for Overweight and Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Collaborators: Westlake University (Other)
Responsible Party: Principal Investigator, Dan Yu, PhD, Principal investigator, Hebei Medical University Third Hospital
Other Study IDs: YD_20190301; NCT07212556 (obsolete NCT alias)
Record Dates: First submitted 2019-12-04; First posted 2019-12-23 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Overweight or Obesity
Keywords: modified Atkins Diet; Overweight; Obesity; Gut Microbiome; Body composition
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, and feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- weight loss group: Dynamic changes in body composition, biochemical metabolomics and gut microbiome will be reported among overweight and obese patients.

SUMMARY:
The aim of the study is to investigate dynamic changes in biochemical metabolism, gut microbiome and its metabolites among overweight and obese participants while they are on a modified Atkins Diets.

DETAILED DESCRIPTION:
The mechanisms of obesity are complex, involved in genes, environment, life style, and systemic and adipose tissue inflammation. Dysbiosis of gut microbiome is considered to make a difference in obesity. On the other hand, both long-term and short-term dietary interventions can induce changes in the body composition and structure and function of gut microbiome. However, it is not really clear how gut microbiome changes along with weight loss in overweight or obese.

In the present study, investigators aim to characterize the gut microbiome among overweight or obese participants on a modified Atkins diets. The stool and blood samples were collected by an interval of every 5% and 10% of weight loss, respectively. Data collecting mainly covers: 1) body composition analysis ; 2) obesity related biochemical metabolism; 3) measurement of gut microbiome using metagenome and 16S rRNA sequencing techniques; 4) metabolomics of serum and gut microbiome; 5) measurement of physical activity and diets using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years old;
2. BMI > 23.9kg/m2;
3. being willing and able to receive guidelines to a modified Atkins diet;
4. signed informed consent.

Exclusion Criteria:

1. patients with serious physical and mental diseases (including cardiovascular and cerebrovascular diseases, liver and kidney diseases, respiratory diseases gastrointestinal diseases, mental diseases, etc.);
2. patients with malignant tumor;
3. pregnant and lactating women;
4. those with recent relocation plans.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study is conducted in Shijiazhuang, a city in Northen China. Eligible participants are residents in this area and aged 18-55 years old, who are on a modified Atkins diet aiming to lose weight.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes of gut microbiome | 36 months
  The stool sample will be collected by an interval of each 5% weight loss that participants experienced. Fecal microbiota will be analyzed by 16S rRNA gene sequencing technique.
Dynamic changes in faecal metabolomics | 36 months
  For participants achieving each 10% weight loss, targeting metabonomics will be applied to identify the abundances of faecal metabolites (e.g. short-chain fatty acids, amino acids and carbohyrates) using validated mass spectrometry methods.

SECONDARY OUTCOMES:
Dynamic changes of body mass index | 36 months
  Weight and height will be combined to report BMI in kg/m^2.
Dynamic changes of body fat | 36 months
  As a body composition parameter, body fat will be analyzed by body composition automatic analyzer for each participant every 10-20 days.
Dynamic changes of muscle mass | 36 months
  Muscle mass will be analyzed by body composition automatic analyzer for each participant every 10-20 days.
Dynamic changes of blood lipids | 36 months
  For participants achieving each 10% weight loss, intravenous serum will be collected and the parameters which can reflect the lipids metalism (such as triglyceride, total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol ) will be measured by automatic biochemical analyzer.
Dynamic changes of fasting blood glucose | 36 months
  For participants achieving each 10% weight loss, intravenous serum will be collected and fasting blood glucose will be measured by automatic biochemical analyzer.
Dynamic changes of homocysteine | 36 months
  For participants achieving each 10% weight loss, intravenous serum will be collected and homocysteine will be measured by automatic biochemical analyzer.
Dynamic changes of blood pressure | 36 months
  For participants achieving each 10% weight loss, blood pressure will be measured by the standard electronic sphygmomanometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Ling Di, MD, Study Director — Hebei Medical University Third Hospital
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
The data might be made available 24 months after completion of the study. Requests for access to the study data can be submitted via email to the principal investigator yudan20122013@163.com, and proposals are required to be attached for approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 24 months after completion of the study
Access Criteria: Qualified researchers engaged in rigorous, independent scientific research; Requests for access to the study data should be submitted via email to the principal investigator yudan20122013@163.com, and proposals are required to be attached for approval.

REFERENCES:
- [Background] Lin BY, Lin WD, Huang CK, Hsin MC, Lin WY, Pryor AD. Changes of gut microbiota between different weight reduction programs. Surg Obes Relat Dis. 2019 May;15(5):749-758. doi: 10.1016/j.soard.2019.01.026. Epub 2019 Jan 31. PMID 30935838
- [Background] Frost F, Storck LJ, Kacprowski T, Gartner S, Ruhlemann M, Bang C, Franke A, Volker U, Aghdassi AA, Steveling A, Mayerle J, Weiss FU, Homuth G, Lerch MM. A structured weight loss program increases gut microbiota phylogenetic diversity and reduces levels of Collinsella in obese type 2 diabetics: A pilot study. PLoS One. 2019 Jul 18;14(7):e0219489. doi: 10.1371/journal.pone.0219489. eCollection 2019. PMID 31318902
- [Background] Heianza Y, Sun D, Smith SR, Bray GA, Sacks FM, Qi L. Changes in Gut Microbiota-Related Metabolites and Long-term Successful Weight Loss in Response to Weight-Loss Diets: The POUNDS Lost Trial. Diabetes Care. 2018 Mar;41(3):413-419. doi: 10.2337/dc17-2108. Epub 2018 Jan 5. PMID 29305401
- [Derived] Yu D, Chen W, Zhang J, Wei L, Qin J, Lei M, Tang H, Wang Y, Xue S, Dong J, Chen Y, Xie L, Di H. Effects of weight loss on bone turnover, inflammatory cytokines, and adipokines in Chinese overweight and obese adults. J Endocrinol Invest. 2022 Sep;45(9):1757-1767. doi: 10.1007/s40618-022-01815-5. Epub 2022 May 30. PMID 35635643